CLINICAL TRIAL: NCT05809427
Title: High Frequency Intraoral Ultrasound Probe for Early Diagnosis of Periodontal Diseases
Acronym: Oralus2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DR220178/ORALUS2; 2022-A01781-42 (Other: IDRCB)
Record Dates: First submitted 2023-03-13; First posted 2023-04-12 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases | interventions — Periodontal Index

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with periodental Disease (Experimental): Imaging/Scanning and recording by Ultrasonic periodontal probing per operator Manual probing per operator with the OMS probe (part of the routine of care)
  Interventions: Device: Periodontal probing

INTERVENTIONS:
Device: Periodontal probing — Imaging/Scanning and recording : Ultrasonic periodontal probing per operator (10 teeth X 6 sites/teeth = 60 probing sites per operator). In addition, 2 teeth per patient will be probed with the ultrasonic probe a second time (2 teeth x 6 sites per tooth = 12 sites per patient) for intra-operator reproducibility purpose.
  Manual probing per operator with the OMS probe (part of the routine of care)

SUMMARY:
The goal of this clinical investigation is evaluation the agreement between the periodontal pocket depth measurement obtained by periodontal probing (gold standard) and the measurement obtained by the ultrasound device

DETAILED DESCRIPTION:
This is a single-center prospective Clinical Investigation in two steps:

Step 1 Preliminary phase : collection and assessment of ultrasonic images to visualize dental and periodontal tissues and structures in order to manually perform periodontal measurements and generate data required for the Artificial Intelligence module training Step 2 : Performance Evaluation : assessment of the ultrasonic probe performance for faster, automatic, accurate and repeatable periodontal measurements in more comfortable conditions for both operator and patient

ELIGIBILITY:
Patient Inclusion Criteria :

Age ≥ 18 years Affiliated to a social security scheme Free, informed and signed consent Ability for participant to comply with the requirements of the study

Exclusion Criteria (patient):

Surgical procedure performed in the area to be scanned Osteosynthesis material Under legal protection Pregnant women, breastfeeding Teeth Inclusion Criteria Minimum of 10 teeth One tooth from each sextant Presence of at least 1/3 of pathological sites (>4mm and/or deep sites >6mm)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2023-07-07 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Periodontal pocket depth measurement by manual probing and measurement by ultrasound probe | 20 minutes for scanning and manual probing
  Periodontal pocket depth measurement by manual probing and measurement by ultrasound probe

SECONDARY OUTCOMES:
Tissues and structures description | 20 minutes for scanning and manual probing(step 1)
  Tissues and structures (alveolar bone, cementum, CEJ, gingiva, enamel) segmentation/labeling and visual identifications on the obtained ultrasonic images
Manual probing measurements with OMS probe (Periodontal pocket depth, Gingival Margin, Clinical Attachment Level) | 20 minutes for scanning and manual probing (step 1)
  Manual probing measurements with OMS probe (Periodontal pocket depth, Gingival Margin, Clinical Attachment Level)
Manual periodontal measurements | 20 minutes for scanning and manual probing](step 1)
  Manunual periodontal measurements (Periodontal pocket depth, Gingival Margin, Clinical Attachment Level) on the ultrasonic images collected and visualized
Patient evaluation questionnaire | 20 minutes for scanning and manual probing (step 2)
  Patient subjective evaluation of the ultrasonic probing protocol (comfort)
Practitioner evaluation questionnaire | 20 minutes for scanning and manual probing (step 2)
  Practitioner subjective evaluation of the ultrasonic probing versus manual probing
Manual probing | 20 minutes for scanning and manual probing (step 2)
  Manual probing with the OMS probe versus Artificial Intelligence (AI) measurements obtained with the ultrasonic probe
The ultrasonic probe measurements performance for intra- operator reproducibility | 20 minutes for scanning and manual probing (step 2)
  Evaluation of the intra-operator reproducibility of the measurements made during ultrasonic probing
Duration of the two exams (Ultrasound scanning versus OMS probe) | 20 minutes for scanning and manual probing (step 2)
  Evaluation of duration of ultrasound scanning and duration of manual probing using a chronometer

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital of Tours, Tours, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Estrade L, Delpierre A, Rimbaud V, Denis F, Rochefort GY, Renaud M. High-frequency intraoral ultrasonography for periodontal tissue characterization: a pilot study exploring echogenic signatures and inflammation detection. BMC Oral Health. 2025 Dec 11;26(1):97. doi: 10.1186/s12903-025-07485-y. PMID 41372763